CLINICAL TRIAL: NCT02939612
Title: Testing a Computerized Interactive Stress Management Intervention in Early Stage Cancer: a Randomized Controlled Trial
Brief Title: Stress Management Intervention in Early Stage Cancer: Randomized Controlled Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Norwegian Cancer Society (Other)
Responsible Party: Principal Investigator, Lise Solberg Nes, Head of Department, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016/1436
Record Dates: First submitted 2016-10-17; First posted 2016-10-20 (Estimated); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Cancer; Stress, Psychological
Keywords: Stress management; App
MeSH Terms: conditions — Neoplasms; Stress, Psychological; Alzheimer Disease | interventions — Amyloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (2):
- App for Stress management (Experimental): Participants will get access to two modules per week for five weeks (total 10 modules). The app consists of stress management education, cognitive behavioral interventions and relaxation training exercises.
  Interventions: Behavioral: App for stress management
- Waitlist control group (No Intervention): Participants will get treatment as usual during the study. After the one year study follow up they will receive the stress management app.

INTERVENTIONS:
Behavioral: App for stress management — An app consisting of 10 modules that teaches stress management, cognitive behavioral coping skills and relaxation training.
  Other Names: Stress management
  Arms: App for Stress management

SUMMARY:
The purpose with this study is to test the effect of an app for stress management among patients with a variety of cancer diagnoses.

DETAILED DESCRIPTION:
A cancer diagnosis and subsequent treatment can be disruptive and traumatic, often accompanied by a multitude of stressors for the patients and their support network. Uncertainty of outcome and invasive medical procedures with aversive side effects are not uncommon, and while people differ widely in how they experience and cope with such challenges, cancer related distress including anxiety, depression, worry and rumination is prevalent. With multiple domains of function impacted it is also not surprising that quality of life (QoL) often is diminished.

Stress management interventions can facilitate adjustment to cancer, including reduced distress and improved quality of life. Unfortunately, many people with cancer do not have the strength or opportunity to attend groups or in-person interventions.

This study will therefore test the effect of an app for stress management among patients with different cancer diagnosis. The app contains 10 modules distributed over five weeks, focusing on education of different techniques for reduction of stress and stress reduction exercises.

The app was tested in a feasibility pilot study among 25 patients with a variety of cancer diagnoses and is now being tested in a randomized controlled trial with a sample of 175 cancer survivors. The participants were randomly assigned to use the 10 module app or to a control group that receive treatment as usual, and will be followed with repeated measures over 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with cancer (all diagnosis).
* Maximum time since completed treatment at hospital: 12 months
* Patients are > 18 years of age, able to write/read/speak Norwegian and have their own smart phone or tablet

Exclusion Criteria:

• None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The Perceived Stress Scale (PSS-14) | Baseline, post intervention follow up at 3, 6, and 12 months
  14 item scale measuring perceived stress. Scale range: 0-56. Higher scores indicate higher perceived stress.

SECONDARY OUTCOMES:
SF-36 Item Short Form Health Survey (RAND-36 version) | Baseline, post intervention follow up at 3, 6, and 12 months
  36 item scale measuring health related quality of life (HRQoL). The scale has 8 subscales and 1 single item score. Scale and single item range: 0 to 100. Higher scores indicate higher HRQoL.
The Self-Regulatory Fatigue-18 (SRF-18) | Baseline, post intervention follow up at 3 and 12 months
  18 item scale measuring self-regulation. Scale range: 18 to 90. A higher score indicates higher self regulatory fatigue
The Brief Coping Orientation to Problems (Brief COPE) | Baseline
  The outcome measure consists of 14 different scales of different coping strategies with two items per scale, for a total of 28 items. Scale range 2 to 8. Higher scores indicate higer use of the different coping strategies
Health, well-being and sleep | Baseline, post intervention follow up at 3, 6, and 12 months
  A 5 item measure, measuring health, well-being and sleep on a scale from 0 to 10. Higher scores indicate better health, well-being and sleep
Intervention commentary | Post intervention (immediately post intervention)
  A six item brief measure of participant's intervention reactions. The first 3 items gauged participants' program perception on a scale from 1 to 5, with 5 indicating better perception. The next 3 items were open ended questions: * What did you like best? * What did you like the least? * Suggestions for improvement?
The Hospital Anxiety and Depression Scale (HADS) | Baseline, post intervention follow up at 3, 6, and 12 months
  14 item scale measuring anxiety and depression. The Scale has a total score with a scale range of 0 to 42 and an anxiety (HADS-A) and a depression (HADS-D) subscale, both with scale range of 0 to 21. Higer scores indicate higher level of anxiety and depression
The Distress Thermometer | Baseline, post intervention follow up at 3, 6, and 12 months
  One item scale measuring distress on a scale from 0 to 10. Higer scores indicate higher distress

CONTACTS AND LOCATIONS:
Overall Officials: Lise Solberg Nes, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Borosund E, Mirkovic J, Clark MM, Ehlers SL, Andrykowski MA, Bergland A, Westeng M, Solberg Nes L. A Stress Management App Intervention for Cancer Survivors: Design, Development, and Usability Testing. JMIR Form Res. 2018 Sep 6;2(2):e19. doi: 10.2196/formative.9954. PMID 30684438